CLINICAL TRIAL: NCT03425227
Title: Frailty Level Monitoring and Analysis After a Pilot Six-week Randomized Controlled Clinical Trial Using FRED Exergame Including Biofeeback Supervision
Brief Title: FRED Exergame Including Biofeeback Supervision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Begoña Garcia Zapirain (Other)
Collaborators: Provincial Council of Bizkaia (Unknown); Basque Government (Unknown)
Responsible Party: Sponsor-Investigator, Begoña Garcia Zapirain, PI of eVIDA Research Group, University of Deusto
Organization: University of Deusto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRED Exergame
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: FRAILTY
Keywords: Frailty; Elderly People; Exergame; Physical Activity; Kinect; Biofeeback
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Blood Pressure; Heart Rate

STUDY DESIGN:
Intervention Model Description: Screening was arranged for 65 subjects in total in accordance with the following criteria.
  Of the 65 individuals who showed interest in taking part in the study, 46 met the inclusion criteria, and these subjects were again asked to carry out some specific tests in order to evidence their degree of frailty.
  Frailty screening was undertaken using the short physical performance battery (SPPB).
  Of the 46 subjects, 40 obtained scores below 10, i.e. 40 subjects may be considered frail.
  In addition to the Barthel scale, the 40 subjects filled in the following questionnaire: EuroQol 5D-5L™. Medical records related to risk of heart failure were also gathered.
  To undertake randomisation, these 40 subjects were classified according to range of age, gender and Barthel score, obtaining a study group and a control group of subjects respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group / control group (Experimental): The subjects belonging to the study group carried out three sessions per week over a 6-week period. Each session involved 20 minutes of activity divided into three parts.
  The subjects belonging to the control group continued to lead their daily lives in the course of which they had no physical activity scheduled.
  Interventions: Other: FRED EXERGAME

INTERVENTIONS:
Other: FRED EXERGAME — biofeedback with physiological constants as follows: systolic blood pressure, diastolic blood pressure, heart rate and blood oxygen saturation
  Other Names: blood pressure, heart rate and blood oxygen saturation were recorded.

SUMMARY:
A pilot six-week randomised controlled trial was carried out introducing biofeedback with physiological constants as follows: systolic blood pressure, diastolic blood pressure, heart rate and blood oxygen saturation in the intervention group.

DETAILED DESCRIPTION:
Objectives:

The main objectives are as follows:

* Verify that the risk of frailty has decreased upon completion of the ExerGame protocol.
* Assess the safety and cardiac healthiness of the exercises done using FRED.

Subject Recruitment Methods:

Contact was established with two residential homes for elderly people, and the necessary permits were requested and obtained from the management at the residential homes.

Approval was requested and obtained from the Ethics Committee in Research of the University of Deusto.

Recruitment at both residential homes was undertaken via informative talks that were given. These talks were open to all interested residents and were advertised via informative posters and pamphlets.

Informed Consent Process:

Interested subjects signed the duly-informed consent form.

Research Procedures:

Screening was arranged for 65 subjects in total in accordance with the following criteria:

Inclusion criteria: persons over 65 years of age with a Barthel score equal to or above 90 points who carry out no scheduled physical activity.

Exclusion criteria: persons over 65 years of age with a Barthel score less than 90 points or with a Barthel score equal to or above 90 points who carry out scheduled physical activity.

Of the 65 individuals who showed interest in taking part in the study, 46 met the inclusion criteria, and these subjects were again asked to carry out some specific tests in order to evidence their degree of frailty.

Frailty screening was undertaken using the short physical performance battery (SPPB), validated and normalised within our milieu, which combines balance testing, gait speed and chair stand. This prioritization was based on its successful validation in detecting frailty and great reliability in predicting disability.

Of the 46 subjects, 40 obtained scores below 10, i.e. 40 subjects may be considered frail.

In addition to the Barthel scale, the 40 subjects filled in the following questionnaire: EuroQol 5D-5L™. Medical records related to risk of heart failure were also gathered.

To undertake randomisation, these 40 subjects were classified according to range of age, gender and Barthel score, obtaining a study group and a control group of subjects respectively.

The subjects belonging to the study group carried out three sessions per week over a 6-week period. Each session involved 20 minutes of activity divided into three parts. The first targeted both the upper and lower extremities, while the second and third targeted specifically the upper and lower extremities respectively. On completion of each part, the subject has the chance to rate the exertion made using the simplified Borg scale [21]. Depending on their rating, they will either be able to continue immediately, or after doing some abdominal-diaphragmatic breathing exercises that will be of a duration that depends on the rating of the exertion made. After completing these breathing exercises, they may choose to continue or otherwise abandon the activity.

The physiological constants - blood pressure, heart rate and blood oxygen saturation - were recorded prior to commencing the FRED game, immediately after completing it and after 5 minutes had elapsed, according to the publications reviewed.

After completing the FRED game session each day, each participant from the study group was asked 2 simple questions, with just a YES or NO answer.

The subjects belonging to the control group continued to lead their daily lives in the course of which they had no physical activity scheduled.

After 6 weeks and having taken part in 18 physical activity sessions with the FRED game, the short physical performance battery (SPPB) test was once again carried out to ascertain whether the degree of frailty had been reduced. The Barthel score and the EuroQol 5D-5L ™ questionnaire were in turn run passed again the subjects and lastly, the system usability scale (SUS) was applied exclusively to subjects from the intervention group.

Instrumentation and Statistical analysis:

FRED is a game developed with the Unity 3D engine. It needs a Kinect game controller connected to a computer and a screen or TV. The measurement of vital signs requires a pulsioxymeter and blood pressure monitor.

For the statistical tests and the creation of graphs, the open-source statistical program R, version 3.2.x for Windows is used.

ELIGIBILITY:
Inclusion Criteria:

* persons over 65 years of age with a Barthel score equal to or above 90 points who carry out no scheduled physical activity.

Exclusion Criteria:

* persons over 65 years of age with a Barthel score less than 90 points or with a Barthel score equal to or above 90 points who carry out scheduled physical activity.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | 10min
  This Battery includes 3 tests: balance test, gait speed and standing up from/sitting down on a chair 5 times. These tests follow a hierarchical sequence.
  A total score is obtained for the whole battery, which is the sum of that obtained from the 3 tests and ranges between 0 and 12, with scores below 10 evidencing frailty.
Barthel Index | 10min
  A scale with which a quantitative estimate is obtained of the degree of independence a subject has to pursue activities of daily living.
  The score ranges 0-100.
EuroQol 5D-5L | 10 min
  A standardised measure for state of health developed by the EuroQol Group in order to provide a single, general measurement applicable to a wide range of health conditions and treatments, which in turn provides a single descriptive profile and a unique state of health rate that may be used in clinical assessment
  . The individual themselves assesses their state of health - first in terms of seriousness via dimensions (descriptive system) and then via a visual analogue scale (VAS) for more general assessment purposes.
The System Usability Scale (SUS) | 10 min
  A questionnaire based on the Likert scale to rate the capacity for using systems.
  The score may be between 0 and 100, in which 100 represents the best usability and a score of ≥68 is considered positive.
Systolic blood pressure | 5 min
  Systolic blood pressure was recorded. Reference value: <150mmHg.
Diastolic blood pressure | 5 min
  Diastolic blood pressure was recorded. Reference value: <90mmHg.
Heart Rate | 2 min
  Heart rate was recorded. Reference value: <76% Maximum heart rate.
Blood Oxygen Saturation | 2 min
  Blood oxygen saturation was recorded. Reference value: Variations <5%SpO2.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Emankor, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Yes
The database will be available at Zenodo.
  Iranzu Mugueta-Aguinaga, & Begonya Garcia-Zapirain. (2018). FRED_DATABASE [Data set]. Zenodo. http://doi.org/10.5281/zenodo.1163736
Time Frame: Until the publication in the journal, the file will be embargoed. After that, the database will be available forever.
Access Criteria: at Zenodo website
URL: http://doi.org/10.5281/zenodo.1163736

REFERENCES:
- [Background] Bouillon K, Kivimaki M, Hamer M, Sabia S, Fransson EI, Singh-Manoux A, Gale CR, Batty GD. Measures of frailty in population-based studies: an overview. BMC Geriatr. 2013 Jun 21;13:64. doi: 10.1186/1471-2318-13-64. PMID 23786540
- [Result] Cabanero-Martinez MJ, Cabrero-Garcia J, Richart-Martinez M, Munoz-Mendoza CL. The Spanish versions of the Barthel index (BI) and the Katz index (KI) of activities of daily living (ADL): a structured review. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):e77-84. doi: 10.1016/j.archger.2008.09.006. Epub 2008 Nov 5. PMID 18990459
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Result] Cabrero-Garcia J, Munoz-Mendoza CL, Cabanero-Martinez MJ, Gonzalez-Llopis L, Ramos-Pichardo JD, Reig-Ferrer A. [Short physical performance battery reference values for patients 70 years-old and over in primary health care]. Aten Primaria. 2012 Sep;44(9):540-8. doi: 10.1016/j.aprim.2012.02.007. Epub 2012 May 16. Spanish. PMID 22608368
- [Result] Freiberger E, de Vreede P, Schoene D, Rydwik E, Mueller V, Frandin K, Hopman-Rock M. Performance-based physical function in older community-dwelling persons: a systematic review of instruments. Age Ageing. 2012 Nov;41(6):712-21. doi: 10.1093/ageing/afs099. Epub 2012 Aug 10. PMID 22885845
- [Result] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Result] O'Brien E, Atkins N, Stergiou G, Karpettas N, Parati G, Asmar R, Imai Y, Wang J, Mengden T, Shennan A; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. European Society of Hypertension International Protocol revision 2010 for the validation of blood pressure measuring devices in adults. Blood Press Monit. 2010 Feb;15(1):23-38. doi: 10.1097/MBP.0b013e3283360e98. No abstract available. PMID 20110786